CLINICAL TRIAL: NCT02588352
Title: Evaluation of Salt Sensitivity in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-01669
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Salts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers (Experimental): Open label administration of salt tablets for one week
  Interventions: Dietary Supplement: Salt tablet

INTERVENTIONS:
Dietary Supplement: Salt tablet — Subjects will be given salt tablets and instructed to take 4 grams of sale three times a day (total of 12 grams of salt/day) for one week

SUMMARY:
The current prospective cross-sectional pilot study is proposed to determine a set of characteristic factors associated with salt sensitivity in young adults by measuring blood pressure, serum aldosterone levels, urine analysis, arterial pulse wave velocity and central arterial pressure in response to short term increases in salt intake.

DETAILED DESCRIPTION:
Since salt sensitivity at an early age is associated with subsequent hypertension and an increase in mortality, intervention by lifestyle modification including the reduction of sodium intake could prevent subsequent increases in blood pressure and development of hypertension, cardiovascular disease and death. It would therefore be beneficial to have a simple method of identifying salt sensitive young adults so that risk factor modification can be achieved to prevent progression of the effects of hypertension on heart function.

This study is a longitudinal pilot study to identify characteristics of salt sensitive young adults so that this population of people can be identified early on and appropriate lifestyle modifications can be made to prevent the subsequent progression of hypertension and cardiovascular disease.

The study will be conducted at 2 visits separated by one week. At the first visit, eligible subjects will be asked to complete questionnaires regarding childhood and current sodium intake.Subjects will be asked about family history of hypertension and cardiovascular disease. Subjects will also undergo blood pressure measurement in both arm, and will provide a blood sample and spot urine sample. Subjects will then be asked to take salt pills 3 times a day for one week, and then return to the study center for a repeat of the above measurements.

ELIGIBILITY:
Inclusion Criteria:

* Young adults age 21-30
* Able and willing to provide written informed consent

Exclusion Criteria:

* Any cardiovascular or other chronic health problem
* Chronic medications besides oral contraceptive pills in women
* BMI>30kg/m2
* Blood pressure >140/90 mmHg
* Inability or unwillingness to adhere to study procedures

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Presence of salt sensitivity | Visit 1 (One Week)
  Defined as an increase in mean arterial blood pressure greater than 5 mmHg

SECONDARY OUTCOMES:
Change in aldosterone level | Baseline to Visit 2 (One Week)
  change in serum aldosterone level
Change in augmentation index (%) | Baseline to Visit 2 (One Week)
  Change in augmentation index determined by radial artery tonometry

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Katz, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be kept on a local server and will be available for sharing based on evaluation of requests from investigators. The transfer of data outside of NYU will be conducted via signed DTA signed by both institutions.